CLINICAL TRIAL: NCT01215240
Title: Prophylactic Peritoneal Dialysis Decreases Time to Achieve a Negative Fluid Balance After the Norwood Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Principal Investigator, Lindsay Ryerson, Clinical assistant professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-LR-001
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome | interventions — Peritoneal Dialysis

STUDY DESIGN:
Intervention Model Description: Subjects randomized to peritoneal dialysis catheter (PDC) or no PDC and standard care.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic peritoneal dialysis (Experimental): Prophylactic peritoneal dialysis
  Interventions: Device: Peritoneal dialysis
- Standard care without PDC (No Intervention)

INTERVENTIONS:
Device: Peritoneal dialysis — Prophylactic peritoneal dialysis
  Arms: Prophylactic peritoneal dialysis

SUMMARY:
Babies born with hypoplastic left heart syndrome (HLHS) have three separate, complex heart surgeries before they turn three years of age. The first surgery typically happens in the first two weeks of life. After this operation, babies come back to the intensive care unit with their chests open. Babies who have heart surgery retain body water after surgery and this extra water slows recovery. Surgeons cannot close the chest until the baby gets rid of the extra water. As a result, babies have to stay in the intensive care unit and on a breathing machine for longer.

Peritoneal dialysis, also known as PD, involves placing a small catheter into the belly cavity at the time of surgery. PD helps the kidney to get rid of extra body water. PD involves putting small amounts of special fluid into the belly through the catheter. This special fluid attracts water and is drained hourly. By allowing the belly cavity to drain, this helps both the heart and the lungs. This allows the chest to be closed and the breathing tube to be removed. The investigators are looking to see how quickly the babies, with and without PD, get rid of the extra water in turn shortening their stay in the intensive care unit and in the hospital. PD is not permanent, and only used for the first few days after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Infants with HLHS or its variants who have a Norwood procedure
* Parental consent

Exclusion Criteria:

* Premature neonates less than 37 weeks gestation
* Weight less than 2 kg
* Urine output less than 0.5ml/kg/hr over 24 hours in the 48 hours prior to the Norwood
* Pre-operative renal replacement therapy
* Abdominal defects precluding placement of a PD catheter
* Known chromosomal abnormality
* Pre-operative cardiopulmonary resuscitation (CPR)
* Pre-operative extra-corporeal life support (ECLS)

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Ryerson, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ryerson LM, Mackie AS, Atallah J, Joffe AR, Rebeyka IM, Ross DB, Adatia I. Prophylactic peritoneal dialysis catheter does not decrease time to achieve a negative fluid balance after the Norwood procedure: a randomized controlled trial. J Thorac Cardiovasc Surg. 2015 Jan;149(1):222-8. doi: 10.1016/j.jtcvs.2014.08.011. Epub 2014 Aug 13. PMID 25218539

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic Peritoneal Dialysis: A peritoneal dialysis catheter (PDC) was inserted at the time of the Norwood operation. The PDC was left open to drainage until the patient was stable enough to start peritoneal dialysis cycles.
  Criteria to start PD cycles included: no fluid bolus given within the past four hours; no escalation of inotropes or vasopressors within the last two hours; vasoactive inotropes score (VIS) ≤ 15; and oxygen saturations ≥ 65% on FiO2 ≤ 0.4.
  PD cycles consisted initially of 10 ml/kg dwell volumes with initial 1.5% dextrose concentration and 60 minute manual cycles (in/dwell 40 minutes, drain 20 minutes).
- Standard Care Without PDC: This group did not receive a peritoneal dialysis catheter at the time of their Norwood. This group received standard care according to their attending physician. At our institution, diuresis is typically initiated with furosemide, either by continuous infusion or bolus dosing at the discretion of the treating team. Study design allowed for placement of a peritoneal dialysis catheter if clinically indicated due to recalcitrant hyperkalemia (serum potassium > 5.9 mEq/L), volume overload unresponsive to diuretics, abdominal compartment syndrome, oliguria (urine output < 1 ml/kg/hr) for more than four hours despite medical intervention or increased serum creatinine in association with persistent metabolic acidosis or low cardiac output syndrome (LCOS).
Period: Overall Study
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Care Without PDC: Standard care with diuretics
- Total: Total of all reporting groups
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: Days] | 9.2 (4) | 9.4 (5.5) | 9.3 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time to First Post-operative Negative 24 Hour Fluid Balance
Description: Time to first post-operative negative fluid balance which occurred in first 72 hrs
Time Frame: up to 72 hours
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Number analyzed (Participants) | 10 | 12
Days | 2.7 (1.06) | 2.67 (0.65)

2. Secondary Outcome: Time to Sternal Closure
Time Frame: Up to 200 hours
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Number analyzed (Participants) | 10 | 12
days | 5.33 (2.87) | 4.17 (1.12)

3. Secondary Outcome: Time to Lactate Less Than or Equal to 2mmol/L
Description: Time to lactate less than or equal to 2mmol/L typically occurred in first 24 hrs
Time Frame: From time of admission in PICU until assessment was reached, assessed up to 24 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Number analyzed (Participants) | 10 | 12
Hours | 15.5 (10.1) | 20.3 (8.3)

4. Secondary Outcome: Time to First Extubation
Time Frame: Up to 15 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Number analyzed (Participants) | 10 | 12
days | 10.1 (4.1) | 8.6 (4.9)

5. Secondary Outcome: Maximum Vasoactive Inotrope Score (VIS) on Post-operative Days 2-5
Description: The maximum VIS assessed from days 2-5 will be chosen. A total VIS score is reported; there are no subscales. Minimum VIS is 0 (there are no units to VIS). Maximum VIS could be 100 but numbers are more typically 5-40. Higher VIS represent more inotropic support and potentially worse outcomes.
Time Frame: Assessed at days 2, 3, 4 and 5 with the highest score from those 4 days reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Number analyzed (Participants) | 10 | 12
score on a scale | 16.4 (9.8) | 15.0 (5.3)

6. Secondary Outcome: Hospital Length of Stay
Time Frame: Assessed up to 8 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
Number analyzed (Participants) | 10 | 12
days | 20.4 (10.8) | 27.7 (21.4)

ADVERSE EVENTS:
Arm/Group | Prophylactic Peritoneal Dialysis | Standard Care Without PDC
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/12
Other Adverse Events (participants affected / at risk) | 6/10 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Peritoneal Dialysis (N=10) | Standard Care Without PDC (N=12)
CPR (Cardiac disorders) | 4 (4) | 0 (0) — Cardiopulmonary resuscitation
ECLS (Cardiac disorders) | 3 (3) | 0 (0) — Extracorporeal life support
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Peritoneal Dialysis (N=10) | Standard Care Without PDC (N=12)
Catheter leakage (Renal and urinary disorders) | 2 (2) | 0
Retention of PD fluid (Renal and urinary disorders) | 4 (4) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No